CLINICAL TRIAL: NCT00005607
Title: A Phase II Study of CPT-11 and 5-FU/LCV in Patients With Previously Untreated Gastric Adenocarcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic or Recurrent Cancer of the Stomach or Esophagus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Robert H. Lurie Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067731; NU-VCCGI9801; P-UPJOHN-976475148; NCI-G00-1740
Record Dates: First submitted 2000-05-02; First posted 2004-08-10 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2000-07

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have metastatic or recurrent cancer of the stomach or esophagus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with metastatic or recurrent adenocarcinoma of the stomach or gastroesophageal junction when treated with irinotecan, fluorouracil, and leucovorin calcium. II. Determine the qualitative and quantitative toxicity, and reversibility of toxicity, of this regimen in this patient population.

OUTLINE: Patients receive irinotecan IV over 90 minutes, leucovorin calcium IV over 15 minutes, and fluorouracil IV once weekly for 4 weeks followed by 2 weeks of rest. Treatment continues every 6 weeks in the absence of unacceptable toxicity or disease progression. Patients are followed at 30 days, and then until death.

PROJECTED ACCRUAL: A total of 18-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or recurrent adenocarcinoma of the stomach or gastroesophageal junction Bidimensionally measurable or evaluable disease Mediastinal or hilar lymph nodes assessed by CT or MRI scan must be at least 2 cm in diameter to be considered measurable Must not be curable with a combination of chemotherapy and radiotherapy No brain metastases No osseous metastasis as only site of disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 3 times upper limit of normal No known Gilbert's syndrome Renal: Creatinine no greater than 1.5 mg/dL Calcium no greater than 12 mg/dL No symptomatic hypercalcemia under treatment Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No history of seizures No serious concurrent infections or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by study complications No psychiatric disorders that would preclude study compliance No other active malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix No uncontrolled diabetes mellitus (i.e., random blood sugar less than 250 mg)

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy for metastatic disease No concurrent immunotherapy Chemotherapy: See Disease Characteristics No prior chemotherapy for metastatic disease No prior radiosensitizing chemotherapy in metastatic setting At least 6 months since prior adjuvant therapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No prior radiotherapy to major bone marrow containing areas (e.g., pelvis, lumbar spine) No prior radiotherapy to only evaluable lesion No concurrent radiotherapy Surgery: At least 1 week since minor surgery and 3 weeks since major surgery and recovered Other: No concurrent phenytoin, phenobarbital, or other antiepileptic prophylaxis No concurrent prochlorperazine on day of irinotecan administration No other concurrent medications except for analgesics, chronic treatments for concurrent medical conditions, or agents required for life threatening medical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02

CONTACTS AND LOCATIONS:
Overall Officials: Al B. Benson, MD, FACP, Study Chair — Robert H. Lurie Cancer Center
Locations (4):
- United States (4):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee